CLINICAL TRIAL: NCT00070668
Title: Inflammatory Genomics in Human Carotid Artery Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1237
Record Dates: First submitted 2003-10-06; First posted 2003-10-09 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Carotid Artery Diseases; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Carotid Artery Diseases; Inflammation

SUMMARY:
To investigate the relationship between genetic variation in genes for inflammation and carotid artery atherosclerosis.

DETAILED DESCRIPTION:
BACKGROUND:

Atherosclerotic vascular disease is a major source of morbidity and mortality. Inflammation plays an important role in atherosclerosis. The tools to systematically study the extent to which genetic variation determines risk of and progression of atherosclerosis are only now becoming available.

DESIGN NARRATIVE:

The study will evaluate the role of genetic variation in inflammatory pathway genes at 29 loci on the risk and progression of carotid artery atherosclerotic disease (CAAD). Genes to be evaluated include those potentially involved in plaque initiation and progression. The investigators will evaluate single nucleotide polymorphisms (SNPs) informative for the common locus haplotypes. Choice of informative polymorphisms for evaluation is based on the genes' evolutionary history. They will evaluate progression effects in subjects with CAAD followed longitudinally by noninvasive magnetic resonance (MR) techniques over 3 years. Risk will be evaluated by case-control comparisons. In additions to evaluating genetic polymorphisms, they will evaluate the intervening phenotypes of protein level for fibrinogen, C-reactive protein, serum amyloid A, and interleukin-6. Independence of genetic predictors from traditional cardiovascular risk factors will be evaluated.

The major specific aims are: Aim 1. Test for inflammatory genetic effects and protein level in CAAD progression in 550 subjects with CAAD (275 with 15-49% and 275 with 50-79% baseline CAAD stenosis) evaluated by 3-year magnetic resonance image follow-up of percent lumen stenosis; Aim 2. Determine whether the variation in the inflammatory genes or protein levels predicts 810 case vs. 810 control status with a case distribution of 335 subject with 15-49%, 275 with 50-75% and 200 with >80% carotid artery stenosis at baseline. Age (onset of vascular disease for cases, current age for controls)-, sex-, race-, and hospital-matched controls will have less than 15% stenosis on carotid duplex ultrasound. Genes that are implicated in disease may eventually allow targeted therapy.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Jarvik — University of Washington